CLINICAL TRIAL: NCT03181737
Title: Psychological Online-training to Optimize Adherence in Patients With Type-II Diabetes a Randomized Controlled Trial (ONSIDE-study)
Brief Title: Psychological Online-training to Optimize Adherence in Patients With Type-II Diabetes
Acronym: ONSIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low adherence rate; need to revise online interventions
Sponsor: Philipps University Marburg (Other)
Collaborators: Prof. Dr. Yvonne Nestoriuc (Unknown); Gaia AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-42k-r
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes mellitus typ 2, adherence, psychological online-intervention, randomized controlled study
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Covivio (Experimental): Covivio is an internet intervention for people with diabetes mellitus type 2. Content is continuously adapted to patients´ concerns and needs. Techniques to promote the disease self-management (i.e. nutrition, exercise), the motivation for health behavior (i.e. discussing pros and cons) conveying goal setting, mediating knowledge about diabetes (i.e. basics, symptoms & complications, diagnosis, therapy) , and reducing depressive symptoms (i.e. increasing activation, mindfulness exercises) are conveyed in interactive sequences that are accompanied by audio recordings, illustrations, and worksheets.
  Patients are also prompted complete brief adherence self-monitoring questionnaires (adherence index) regularly. Optional text messages with motivational content accompany the program daily. The program can be accessed for 56 days after registration.
  Interventions: Behavioral: Covivio/Relaxio
- Relaxio (Active Comparator): Relaxio is a psychological online-relaxation-training. The purpose of the program is to improve the self-management of diabetes by relaxation and stress reduction. The program consist of three types of exercises (1) imagination (i.e. sunset, mountain lake), (2) breathing techniques (i.e. balancing, calm breathing), and (3) body exercises (i.e. relaxing body journey, progressive muscle relaxation (PMR)). The exercises are supported by audio files (optionally also for reading). Optional weekly text messages with motivational content accompany the program. The program can be accessed for 56 days after registration.
  Interventions: Behavioral: Covivio/Relaxio
- Care-as-Usual (CAU) / wait list (No Intervention): In the CAU/wait list control group, participants are free to continue to engage with any treatment they require (i.e., CAU). However, they will receive access to Covivio six months post-baseline (i.e., wait list with respect to Covivio access).

INTERVENTIONS:
Behavioral: Covivio/Relaxio — Informations already included in arm/group descriptions.
  Arms: Covivio; Relaxio

SUMMARY:
The trial aim of the study is to evaluate the effectiveness of a novel psychological internet intervention (Covivio), which was designed to improve adherence in Persons with Diabetes Mellitus type 2 (PwDM), using cognitive-behavioral therapy (CBT) techniques. Therefore, 300 PwDM will be recruited and randomized to three groups:

(1) a treatment group that immediately receives two-month access to Covivio and may also use care-as-usual (CAU), (2) an active control group that also immediately receives a two-month access to Relaxio, an internet program with the focus of stress relaxation ,and may also additionally use CAU or (3) a control group, in which they may engage with any diabetes treatment (i.e. CAU/ wait list control group). The active control group (2) and the wait control group (3) receive access to Covivio after a delay of six months. The primary outcome measure is the Diabetes Self-Management Questionnaire-Revised (DSMQ-R), collected at baseline, two (post-treatment), and additionally three and six months follow-up.

DETAILED DESCRIPTION:
The treatment of diabetes type 2 is a major challenge for the health care system. According to the International Diabetes Federation (IDF), around 382 million people between the ages of 20 and 79 are currently affected worldwide. The presence of diabetes is associated with personal suffering, impaired quality of life and a deficient treatment leads to complications like retinal ablation, neuropathy, nephropathy and the diabetic-foot syndrome. An appropriate treatment is dedicated to the purpose of adjusting the blood glucose, is very complex and involves many areas of life. Internet-administrated psychological interventions are easily accessible and preliminary evidence suggests that online programs promote lifestyle changes, i.e. nutrition and exercises, of people with diabetes mellitus type 2. However, no trial has yet examined weather a CBT-based internet intervention designed to meet the needs of PwDM can achieve sustained improve adherence behavior like nutrition, physical activity and medication intake, when offered as adjunct to treatment as usual.

The internet-based intervention evaluated in this trial was designed with the aim of enhancing adherence to PwDM over a period of 60 days. The intervention focuses issues in disease self-management including lifestyle habits (e.g. nutrition, exercise) and medication adherence. The program comprised psychotherapeutic techniques gleaned primarily from CBT to promote motivation for health behavior, conveying goal setting, mediating knowledge about diabetes (basics, symptoms & complications, diagnosis, therapy) , and increasing activation to reduce depressive symptoms and increasing mindfulness skills. The delivery and training of content is continuously individualized to match users' preferences and needs, based on responses within the program. The intervention is delivered via the Internet and protected by individually assigned passwords.

This randomized controlled trial will include 300 participants with diabetes mellitus type 2. Participants will be recruited from various settings, including diabetes outpatient treatment centers and internet forums/groups. Methods such as newspaper articles, flyers, posters, and media articles will be used to inform potential participants about the study (all material will be in German). Participants will be screened for inclusion and exclusion criteria via telephone, and randomly assigned to either (1) a treatment group that may use care as usual (CAU) and in addition immediately receives two-month access to the novel, internet -administrated intervention (Covivio), (2) an active control group that may also use CAU and in addition immediate receives two-month access to a psychological online-relaxation-training (Relaxio), or (3) a wait list control group, in which they receive CAU. Measurements are collected online at pre-treatment (T0), post-treatment (T1), and three (T2) and six months (T3) follow-up. After the last follow-up (T3), all participants gain access to the online-program which they had not yet been able to use.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Diagnosis of type 2 diabetes mellitus (T2DM) and HbA1c > 6,5%;
* currently deficient self-management behavior, as operationalized by a score of less then 7,5 on the DSMQ-R
* Regular control (every 3 months) of the HbA1c by physicians during the study period
* ability to speak and read German
* access to the internet and personal possession of an appropriate device on which the internet-based intervention can be used regularly (e.g., smartphone, computer, laptop)
* expressed motivation to participate in the trial and use an internet-based intervention to acquire skills and knowledge that may aid in the treatment of diabetes mellitus

Exclusion Criteria:

* other known major mental disorder, such as bipolar disorder, schizophrenia or another psychotic disorder, or borderline personality disorder (based on the MINI interview) or acute and serve physical disease
* acute suicidality (that is, intention or plan to commit suicide, as assessed with the respective module of the MINI interview)
* newly prescribed diabetes medication or change in diabetes medication dosage in month prior to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Management Questionnaire (DSMQ-R) | Changes from baseline to 2, 5 and 8 months post-baseline.
  Self-report of diabetes self-management , to measure adherence to diabetes treatment. Diabetes self-management behavior with a focus on behavioral patterns which contribute to a stable blood glucose level (nutrition, medication adherence, blood glucose self-monitoring, exercise, regular medical examinations).

SECONDARY OUTCOMES:
Glycemic control | Change from baseline in HbA1c level to 3 months (also assessed at 6 months post baseline)
  Change in participant's HbA1c level
GLTEQ (Godin- Leisure- Time Exercise Questionnaire) | changes from baseline to 2 months (also assessed at 5 and 8 months post baseline)
  Self-report measure of leisure-time exercise habits
PAID (Polonsky, Problem Areas in Diabetes Questionnaire) | Changes from baseline to 2 months (also assessed at 5 and 8 months post baseline)
  Self-report measure of diabetes specific strains
GAD-7 (Generalized Anxiety Disorder Assessment) | Changes from baseline to 2 months (also assessed at 5 and 8 months post baseline)
  Self-report anxiety symptom severity measure
PHQ-9 (Patient Health Questionnaire) | Changes from baseline to 2 months (also assessed at 5 and 8 months post baseline)
  Self-report measure of depressive symptoms
WHO-5 (WHO-Five Well-Being Index) | Changes from baseline to 2 months (also assessed at 5 and 8 months post baseline)
  Self-report measure of general well-being
Subjective usefulness of the program | Assessed at 2 months post baseline
  Individually designed self-report items

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, Philipps University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data shall be made available upon request for projects such as meta-analyses after completion of the study